CLINICAL TRIAL: NCT05168683
Title: A Phase 1, Single Centre, Two-Part, Open Label, Crossover Study in Healthy Volunteers Using Scintigraphy to Characterize the In Vivo Performance of ALLN-346 Enteric Coated Tablets
Brief Title: Scintigraphy Study in Healthy Volunteers to Characterize the Performance of ALLN-346 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allena Pharmaceuticals (Industry)
Collaborators: BDD Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ALLN-346-103
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Hyperuricemia; Gout
MeSH Terms: conditions — Hyperuricemia; Gout

STUDY DESIGN:
Intervention Model Description: Subjects in each study Part participate in all treatment arms of that Part.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part One (Experimental): Four Study Treatments will be dosed during Part One of the study with radiolabelled ALLN-346 tablets (in 12 subjects): Treatment A ALLN-346 enteric coated (EC) fast release tablet; Treatment B ALLN-346 fast release capsule; Treatment C ALLN-346 EC slow release tablet; Treatment D ALLN-346 slow release capsule. Subjects will be dosed in a lightly fed state.
  Interventions: Drug: Each ALLN-346 treatment will be radiolabelled to contain 4 MBq 99mTc at time of dosing with light meal
- Part Two (Experimental): Following completion of Part One of the study, study treatment (one or both of those administered in Part One) and dosing requirements will be confirmed for dosing in Part Two, to be administered in fasted and/or fed states (in 12 subjects).
  Interventions: Drug: Each ALLN-346 treatment will be radiolabelled to contain 4 MBq 99mTc at time of dosing in fasted/fed state

INTERVENTIONS:
Drug: Each ALLN-346 treatment will be radiolabelled to contain 4 MBq 99mTc at time of dosing with light meal — Dosing or radiolabelled ALLN-346 fast or slow release tablets or capsules. Scintigraphic images will be taken
  Other Names: Engineered urate oxidase radiolabelled
  Arms: Part One
Drug: Each ALLN-346 treatment will be radiolabelled to contain 4 MBq 99mTc at time of dosing in fasted/fed state — Selected dosing of Part One treatments in fasted and/or fed states
  Other Names: Engineered urate oxidase radiolabelled
  Arms: Part Two

SUMMARY:
The purpose of the study is to understand the gastrointestinal transit time and disintegration behavior of the formulations in vivo in normal healthy volunteers when ALLN-346 formulations are given with light meal or in fasted or other fed states.

DETAILED DESCRIPTION:
This study includes two parts. Part One will evaluate two ALLN-346 formulations, a fast release and a slower sustained release. Subjects will receive a single tablet of each formulation and a capsule of each formulation at separate assessment visits. Subjects will attend a maximum of 4 assessment visits. The primary purpose of this part of the study is to understand the gastrointestinal transit time and disintegration behaviour of the formulations in vivo in normal healthy volunteers when ALLN-346 formulations are given with light meal.

Part Two will involve a second cohort of subjects and will comprise further scintigraphic studies on one or both formulation(s) from Part One in fasted and/or fed states. Subjects will attend a maximum of 4 assessment visits, the number of treatment arms will be decided following completion of Part One.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 30 kg/m², inclusive.
* Body weight ≥50 kg
* Voluntary written informed consent
* Good general health with no clinically significant and/or relevant abnormalities of medical history or prior to dosing evaluations, including physical examination, vital signs and ECG and screening clinical laboratory results

Exclusion Criteria:

* Current or recurrent disease that could affect the study conduct or laboratory assessments
* History of current or relevant previous non-self-limiting gastrointestinal disorders
* Currently suffering from disease known to impact gastric emptying, e.g., migraine, Type 1 or Type 2 diabetes mellitus
* Untreated hypertension or has hypertension under treatment.
* Diagnosis of an immunosuppressive illness or a condition requiring chronic immunosuppression.
* As a result of a physical examination or screening investigations, and available prior to dosing evaluations, the PMI or medically qualified designee/physician responsible considers the volunteer unfit for the study
* Any contradictions to the gamma scintigraphy procedure
* Measured body temperature >38°C at screening visit (COVID-19 risk reduction procedure)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Scintigraphic images to detect transit time of radiolabel release | 12 hours
  To assess the onset of disintegration/release with transit time for the radiolabelled study treatments in each ALLN-346 formulation

SECONDARY OUTCOMES:
Incidence of Adverse Events | 14 Days
  Number of subjects with treatment emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christine Tosone, Study Director — Allena Pharmaceuticals, Inc.
Locations (1):
- BDD Pharma Ltd Bio-Imaging Centre Within Glasgow Royal Infirmary, Glasgow, Scotland, United Kingdom